CLINICAL TRIAL: NCT01847625
Title: Safe Traction During Ongoing Lead Extraction Procedure
Brief Title: Safe Traction During Ongoing Lead Extraction Procedure (STOP)
Acronym: STOP
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-011
Record Dates: First submitted 2013-04-09; First posted 2013-05-07 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Electrode Malfunction; Infections of Cardiac Electronic Implantable Devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physicians experienced in lead extraction: Physicians experienced in lead extraction
  Interventions: Other: simulator

INTERVENTIONS:
Other: simulator

SUMMARY:
The study will evaluate (in-vitro) the forces that are typically used for the extraction of pacemaker or defibrillator electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Experience in pacemaker and defibrillator lead extraction

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians experienced in pacemaker or defibrillator electrode extraction
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Forces used for lead extraction | 10 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany

REFERENCES:
- [Result] Lennerz C, Pavaci H, Grebmer C, von Olshausen G, Semmler V, Buiatti A, Reents T, Ammar S, Deisenhofer I, Kolb C. Forces applied during transvenous implantable cardioverter defibrillator lead removal. Biomed Res Int. 2014;2014:183483. doi: 10.1155/2014/183483. Epub 2014 May 21. PMID 24967337